CLINICAL TRIAL: NCT03972384
Title: A Problem Solving Intervention for Post-ICU Cognitive Impairment in Older Adults
Acronym: PIC-UPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Judith Tate, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019H0089
Record Dates: First submitted 2019-04-08; First posted 2019-06-03 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Critical Illness; Mechanical Ventilation Complication; Delirium; Cognitive Impairment
Keywords: Post-ICU Syndrome; Recovery; Home Discharge; Problem Solving; Adaptation
MeSH Terms: conditions — Critical Illness; Delirium; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two groups randomized to treatment (Post-ICU problem solving program) or usual care (no Post-ICU problem solving program).
Who Masked: Outcomes Assessor
Masking Description: Data collectors are blind to condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-ICU Problem Solving (Experimental): The PIC-UPS intervention focuses on self-regulation activities and environmental cues to overcome problems with memory, planning and decision-making. The interventionist uses guided discovery, reviews progress, and emphasizes generalization and transfer to other patient-identified problems. This approach may be more acceptable to participants because they can see the relevance of tasks to everyday life. Activities such as goal-setting, self-evaluation and reflective thinking behaviors enhance self-efficacy and increase the likelihood that the individual will engage in self-management behaviors. The first session of PIC-UPS will be delivered after enrollment to those participants randomized to the intervention group. Weekly intervention sessions will be conducted by a trained interventionist and supplemented by telephone reminders to complete daily homework. Follow-up data collection will be conducted in the home by a blinded data collector three months post-enrollment.
  Interventions: Behavioral: Post-ICU Problem Solving
- Control Group (No Intervention): Participants in the control group will complete several surveys upon enrollment and randomization. Follow-up data collection will be conducted in the home for all participants control group by a blinded data collector three months post-enrollment.

INTERVENTIONS:
Behavioral: Post-ICU Problem Solving — We have adapted the Cognitive Orientation to Daily Occupational Performance (CO-OP) as the Post-ICU Problem Solving intervention to be delivered in the home to patients following an illness that required an ICU stay. CO-OP is a form of meta-cognitive strategy training that teaches individuals to identify and prioritize problematic daily activities, identify barriers impeding performance, generate and evaluate strategies addressing these barriers, and generalize learning through practice. Thus, strategy training teaches skills that can be used to address disability in "real-life" activities, and is integral to personalized rehabilitation services. CO-OP has been adapted in numerous settings and most recently, it is being utilized successfully in patients with acquired cognitive dysfunction following acute stroke. This represents a useful intervention, tested in similar populations with minimal risk to the participants and potential for maximal benefit for this population.
  Other Names: PIC-UPS
  Arms: Post-ICU Problem Solving

SUMMARY:
This study will apply an evidence based program to assist ICU survivors to overcome cognitive problems as a result of their critical illness. This study will determine feasibility of recruitment, retention and engagement with the program as well as acceptability of the program to the participants.

DETAILED DESCRIPTION:
The Post-Intensive Care Unit Problem Solving (PIC-UPS) is an adaptation of a problem solving strategy developed and tested in diverse patient populations. Its effectiveness has been demonstrated in children with movement disorders or learning difficulties as well as adults with cognitive problems following acute stroke. Participants will be randomized onto usual care and intervention groups. The usual care group will complete study surveys after enrollment and 10 weeks after enrollment. The intervention group will receive the following: In the (PIC-UPS) program, participants will be engaged for 10 sessions, learning how to do skills they select as treatment goals. The first session consists of an assessment, and selecting the goals to meet during the 10 sessions. In the next sessions, conducted at the participant's home, participants practice the skills selected as treatment goals, and assisted by the study team, use strategies to help better learn and perform those skills. Some examples of tasks that others have addressed in these sessions are gardening, yoga breathing, handwriting, managing family finances, medication management, or initiating an exercise regimen. Participants will be encouraged to select tasks most relevant and problematic to their unique situation. In addition to attending the sessions, the participants will be asked to rate the sessions and asked about how useful they were in helping to achieve goals. This involves the completion of some written questionnaires and will take about a half hour.

Sample Assessment and Treatment Schedule Session Description

1. Assessment session approximately one and a half hours long. Combination of questionnaires and goal setting interview. Baseline testing of 3 goals.
2. Treatment session + 2 surveys, approximately one hour long.
3. Treatment session 3, approximately one hour long.
4. Treatment session 4, approximately one hour long.
5. Treatment session 5, approximately one hour long.
6. Treatment session 6, approximately one hour long.
7. Treatment session 7, approximately one hour long.
8. Treatment session 8, approximately one hour long.
9. Treatment session 9, approximately one hour long.
10. Treatment session 10, followed by first post-intervention assessments, approximately 2 hours long.

ELIGIBILITY:
Inclusion Criteria:

* >55 years old
* discharged home following an ICU stay,
* reside at home and were functionally independent prior to admission to the ICU based on family report,
* speak and read English,
* mechanically ventilated for at least 48 hours,
* have more than one positive clinical measurement of delirium during the ICU stay,
* Montreal Cognitive Assessment score (MoCA) between 25-17.

Exclusion Criteria:

* Pre-illness diagnosis of dementia or pre-morbid cognitive impairment (IQCODE score >3.51);
* profound uncorrected visual or hearing impairment that precludes use of the telephone;
* psychiatric condition that precludes full participation in the intervention;
* substance abuse as measured by cut-off score of 2 on CAGE-Substance Abuse Screening Tool;
* discharge to hospice care.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change of Cognitive function as measured by Self-Administered Gerocognitive Examination | Week 1 and week 12
  Measure of the program's effect on Cognitive Function as measured using the Self-Administered Gerocognitive examination (SAGE) The maximum score is 22. A score of 17 and above is considered normal.
Change in development of Chronic Illness self management practices(as measured by Self-Efficacy Scale) | Week 2 and Week 12
  Determine the program's effect on Chronic Illness self- management as measured by the Self-Efficacy to Manage Chronic Disease Scale which is made up of 6-items on a visual analog scale, ranging from 1 (not at all confident) to 10 (totally confident).
Change in medication adherence practices (as measured by Medication Management Instrument for Deficiencies in the Elderly (MedMaIDE)) | Week 2 and Week 12
  Measure change in medication Adherence by using the MedMaIDE scale that contains a maximum total score of 13.
Change in participant's rate of depression as measured by Patient Health Questionnaire - 2) | Week 1 and Week 12
  Measure of the program's effect on rate of depression
Change in anxiety levels as measured by Geriatric Anxiety Scale (GAS) | Week 1 and Week 12
  Measure change in participant's anxiety levels as measured by Geriatric Anxiety Scale that contains 10 questions on anxiety with a scoring scale of 1-6 = Minimal; 7-9 = Mild, 10 = Moderate; 12-30 = Severe.
Change in depression levels as measured by Geriatric Depression Scale (GDS) | Week 1 and Week 12
  Measure change in participant's depression levels as measured by Geriatric Depression Scale that contains 15 questions on depression. A score of 5 or more suggests depression.
Change in Health related Quality of Life by a Short Form Health Survey - 36 | Week 1 and Week 12
  Measures Health Related Quality of Life
Assess the effect of the Post-Intensive Care Problem Solving program through intervention completion rates | 15 months
  Assess the effect of the Post-intensive care program through intervention completion rates.
Access change in participant use of the health system | Week 12
  Access change in frequency of use of health system by use of the health system by number of times the study participatns use emergency department services, phone calls to physicians.
Assess change in functional independence when performing activities of daily living as measured by the Katz Activities of Daily Living Scale. | Week 1 and Week 12
  Measure change in participant's functional independence when performing activities of daily living using the Katz Activities of Daily Living Scale. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Assess change in functional independence when performing instrumental activities of daily living using the Lawton Instrumental Activities of Daily Living. | Week 1 and Week 12
  Assess changes in functional independence when performing instrumental activities of daily living using the Lawton Instrumental Activities of Daily Living. There are eight domains of function measured with the Lawton IADL scale.
  Women are scored on all 8 areas of function; historically, for men, the areas of food preparation, housekeeping, laundering are excluded.
  Clients are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Tate, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No